CLINICAL TRIAL: NCT05119049
Title: Efficacy of Aquatic Physiotherapy in the Treatment of Upper Limb Lymphedema in Women With Breast Cancer: a Randomised Controlled Trial.
Brief Title: Efficacy of Aquatic Physiotherapy in the Treatment of Upper Limb Lymphedema in Women With Breast Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isabel Lopez Zamora (Other)
Responsible Party: Sponsor-Investigator, Isabel Lopez Zamora, Physiotherapist, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILZamora
Record Dates: First submitted 2021-10-23; First posted 2021-11-12 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: Experimental study randomized controlled
Who Masked: Investigator
Masking Description: The initial, intermediate and final evaluations were carried out by a blind researcher, not familiar with the group assigned to the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic exercise plan in the pool. (Experimental): The experimental group underwent 20 sessions with an aquatic exercise plan in the pool at the rehabilitation department.
  Interventions: Other: Exercise guideline
- Exercises in a rehabilitation room. (Active Comparator): The control group did the same exercises and sessions in one of the rooms in the rehabilitation department.
  Interventions: Other: Exercise guideline

INTERVENTIONS:
Other: Exercise guideline — The experimental group underwent 20 sessions with an aquatic exercise plan in the pool at the rehabilitation department. The control group did the same exercises in one of the rooms in the rehabilitation department, with the same number of sessions. Both groups were guided by a physiotherapist. The main outcome variables were assessed at the start of the study, at the end of the 20 sessions, and at 3 months after completing the sessions.

SUMMARY:
This study aims to evaluate the effectiveness of Aquatic Therapeutic Exercise by providing a set of exercises in the reduction and / or control the volume of secondary lymphedema treatment of breast cancer in patients who are in the maintenance phase of conventional treatment. It is an experimental, randomized, unifactorial, and intersubjective study. The intervention group will be treated by guided underwater exercises while the control group will receive the same set of exercises out-of-water. The research will be based on comparing the difference on the volume of lymphedema obtained by the exercises provided aquatic environment and out-of-water exercises. The study population will be obtained from rehabilitation service Bellvitge Hospital. The goal is to evaluate the volume of lymphedema and the quality of life related to the health of patients will be evaluated before starting the treatment, at the end of the 20 sessions, when the treatment reaches 3 months and when patient is discharged.

DETAILED DESCRIPTION:
A randomized controlled experimental study has been carried out where two work groups were compared, experimental N: 43 that carried out an exercise regimen designed in the aquatic environment and control N: 47 that carried out the same regimen of exercises in a physiotherapy room. Both groups did 20 treatment sessions of 45 minutes duration with a frequency of 2 or 3 days per week. Lymphedema changes, quality of life and adherence to treatment were evaluated. The evaluations were 3 days prior to the start of the program, at the end of the 20 sessions, and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Female gender.
* Age between 18 and 75 years.
* Diagnosis of lymphedema in the upper limb secondary to breast cancer treatment.
* Present mild lymphedema or moderate (types I and II respectively according to the volumetric classification of the types of edema according to severity).

Exclusion Criteria:

* Primary lymphedema or secondary to other surgery.
* Bilateral lymphedema.
* Presence of hydrophobia.
* Severe cardiovascular and respiratory diseases.
* Urinary and fecal incontinence.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 90 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Volume of the affected limb. | 3 days before the start of the program, at 30 days, and at 3 months after completing the sessions.
  The investigators assessed changes in the volume of the affected limb over a specified period of time and possible long-term improvements. The independent variable studied was the effect of exercise in water compared with exercise out of water.
  The expected outcome (dependent variable) was a reduction or maintenance of the volume of the lymphedema-affected limb. A measuring tape was used to take serial circumferential measurements of both limbs using anatomical reference points on both sides.

SECONDARY OUTCOMES:
Quality of life health related. | 3 days before the start of the program, at 30 days and at 3 months after completing the sessions.
  FACT-B+4 scale: general physical wellbeing, family/social wellbeing, emotional wellbeing, functional wellbeing and additional patient concerns.
Adherence | At 3 months after completing the sessions.
  Rate of adherence to treatment. Adherence to treatment questionnaire: YES / NO
Age. | 3 days before the start of the program.
  Possible influence of age and confounding factors.
Severity of lymphedema | 3 days before the start of the program, at 30 days and at 3 months after completing the sessions.
  Volume of limb. Possible influence and confounding factors.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel López Zamora, physiotherapist, Principal Investigator — Bellvitge Hospital

IPD SHARING:
Plan to Share IPD: No